CLINICAL TRIAL: NCT04483739
Title: Phase III Study of Isatuximab-Carfilzomib-Lenalidomide-Dexamethasone (Isa-KRd) Versus Carfilzomib-Lenalidomide-Dexamethasone (KRd) in Newly Diagnosed Multiple Myeloma Patients Eligible for Autologous Stem Cell Transplantation (IsKia TRIAL
Brief Title: Isa-KRd vs KRd in Newly Diagnosed Multiple Myeloma Patients Eligible for Autologous Stem Cell Transplantation (IsKia TRIAL)
Acronym: IsKia
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: EMN Trial Office S.r.l. Impresa Sociale (Other); Sanofi (Industry); Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMN24
Record Dates: First submitted 2020-06-23; First posted 2020-07-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
Keywords: newly diagnosed MM; autologous stem cell transplantation; Isatuximab; Carfilzomib; Lenalidomide; Dexamethasone
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Krd Induction (Experimental): 4 28 day cycles of Carfilzomib = 20 mg/m2 IV on day 1 cycle 1 only, followed by 56 mg/m2 IV on days 8, 15 cycle 1 and on days 1, 8, 15 for cycles 2-4 Lenalidomide= 25 mg orally daily on days 1-21 Dexamethasone = 40 mg orally/IV on days 1, 8, 15, 22
  Interventions: Drug: Carfilzomib Lenalidomide Dexamethasone
- Isa-KRd induction (Experimental): Isatuximab= 10 mg/kg IV on day 1, 8, 15, and 22 during Cycle 1, followed by 10 mg/kg IV on days 1 and 15 during Cycles 2 to 4.
  Carfilzomib = 20 mg/m2 IV on day 1 cycle 1 only, followed by 56 mg/m2 IV on days 8, 15 cycle 1 and on days 1, 8, 15 for cycles 2-4 Lenalidomide= 25 mg orally daily on days 1-21 Dexamethasone = 40 mg orally/IV on days 1, 8, 15, 22
  Interventions: Drug: Isatuximab Carfilzomib Lenalidomide Dexamethasone
- KRd post ASCT consolidation (Experimental): 4 28 day cycles of Carfilzomib = 56 mg/m2 IV on days 1, 8, 15 cycle 5-8 Lenalidomide= 25 mg orally daily on days 1-21 Dexamethasone = 40 mg orally/IV on days 1, 8, 15, 22
  Interventions: Drug: Carfilzomib Lenalidomide Dexamethasone
- Isa-KRd post ASCT consolidation: (Experimental): 4 28 day cycles of Isatuximab= 10 mg/kg IV on days 1 and 15 on cycles 5-8 Carfilzomib = 56 mg/m2 IV on days 1, 8, 15 cycle 5-8 Lenalidomide= 25 mg orally daily on days 1-21 Dexamethasone = 40 mg orally/IV on days 1, 8, 15, 22
  Interventions: Drug: Isatuximab Carfilzomib Lenalidomide Dexamethasone
- KRd light consolidation (Experimental): 12 28 day cycles of Carfilzomib = 56 mg/m2 IV on days 1, 15 Lenalidomide = 10 mg orally on days 1-21 Dexamethasone = 20 mg orally/IV on days 1, 15
  Interventions: Drug: Carfilzomib Lenalidomide Dexamethasone
- Isa-KRd light consolidation (Experimental): Isatuximab= 10 mg/kg IV on day 1 Carfilzomib = 56 mg/m2 IV on days 1, 15 Lenalidomide = 10 mg orally on days 1-21 Dexamethasone = 20 mg orally/IV on days 1, 15
  Interventions: Drug: Isatuximab Carfilzomib Lenalidomide Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib Lenalidomide Dexamethasone — Isatuximab-Carfilzomib-Lenalidomide-Dexamethasone (Isa-KRd) versus Carfilzomib-Lenalidomide-Dexamethasone (KRd) in newly diagnosed multiple myeloma patients eligible for autologous stem cell transplantation
  Other Names: KRd
  Arms: KRd light consolidation; KRd post ASCT consolidation; Krd Induction
Drug: Isatuximab Carfilzomib Lenalidomide Dexamethasone — Isatuximab-Carfilzomib-Lenalidomide-Dexamethasone (Isa-KRd) versus Carfilzomib-Lenalidomide-Dexamethasone (KRd) in newly diagnosed multiple myeloma patients eligible for autologous stem cell transplantation
  Other Names: Isa-KRD
  Arms: Isa-KRd induction; Isa-KRd light consolidation; Isa-KRd post ASCT consolidation:

SUMMARY:
This protocol is a phase III study designed to compare the efficacy and the safety of Isa-KRd induction, transplant, Isa-KRd post ASCT consolidation and Isa-KRd light consolidation vs KRd induction, transplant, KRd post ASCT consolidation and KRd light consolidation After confirmation of eligibility criteria patients will be randomized to one of the 2 treatment groups in a 1:1 randomization ratio.

DETAILED DESCRIPTION:
This is a open-label randomized phase III study that enrolls newly diagnosed MM patient eligible for high-dose chemotherapy and ASCT. Patients will be randomized at enrolment (1:1, stratification according to ISS Stage [3 levels: I vs II vs III] and cytogenetic risk FISH [2 levels: high-risk vs standard risk/missing] based on presence of t(4;14), t(14;16), and/or del 17p)) into 2 treatment arms: -ARM A: induction with 4 cycles of Isatuximab-Carfilzomib-Lenalidomide-dexamethasone (Isa-KRd) followed by cyclophophamide and stem cell collections, chemotherapy with Melphalan 200 mg/m2 followed by ASCT (Mel200-ASCT), 4 cycles of Isa-KRd post ASCT consolidation and 12 cycles of Isatuximab-Lenalidomide-Carfilzomib-dexamethasone (IsaKRd) light consolidation; ARM B: induction with 4 cycles of Carfilzomib-Lenalidomide-dexamethasone (KRd) followed by cyclophophamide and stem cell collections, chemotherapy with Melphalan 200 mg/m2 followed by ASCT (Mel200-ASCT), 4 cycles of KRd post ASCT consolidation and 12 cycles of Carfilzomib-Lenalidomide-dexamethasone (KRd) light consolidation. Details of all treatments (dose and schedule) are given in paragraph 8. After light consolidation patients are allowed to receive Lenalidomide maintenance as per standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patient with newly diagnosed multiple myeloma and eligible to ASCT.
* Patient is, in the investigator's opinion, willing and able to comply with the study visits and procedures required per protocol.
* Patient has provided written informed consent in accordance with federal, local, and institutional guidelines prior to initiation of any study-specific activities or procedures. Subject does not have kind of condition that, in the opinion of the Investigator, may compromise the ability of the subject to give written informed consent and patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Monoclonal plasma cells in the bone marrow ≥10% or presence of a biopsy proven plasmacytoma and documented multiple myeloma satisfying at least one of the calcium, renal, anemia, bone (CRAB) criteria or biomarkers of malignancy criteria:
* CRAB criteria:

  * Hypercalcemia: serum calcium >0.25 mmol/L (>1 mg/dL) higher than upper limit of normal (ULN) or >2.75 mmol/L (>11 mg/dL)
  * Renal insufficiency: creatinine clearance <40mL/min or serum creatinine >177 μmol/L (>2 mg/dL)
  * Anemia: hemoglobin >2 g/dL below the lower limit of normal or hemoglobin <10 g/dL
  * Bone lesions: one or more osteolytic lesions on skeletal radiography, CT, or PET-CT
* Biomarkers of Malignancy:

  * Clonal bone marrow plasma cell percentage ≥60%
  * Involved: uninvolved serum FLC ratio ≥100
  * >1 focal lesion on magnetic resonance imaging (MRI) studies
* Patient is 18 - 70 years old and is eligible for autologous stem cell transplantation
* Patient has measurable disease as defined by any one of the following:

  * Serum monoclonal paraprotein (M-protein) level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours; or
  * Light chain multiple myeloma without measurable disease in the serum or the urine: Serum immunoglobulin FLC ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda FLC ratio.
* Life expectancy ≥ 3 months
* ECOG status ≤2
* Clinical laboratory values meeting the following criteria during the Screening Phase:

  * Adequate hepatic function, with serum (alanine aminotransferase) ALT ≤ 2.5 times the upper limit of normal (ULN), AST (aspartate transaminase) ≤ 2.5 x the ULN
  * Serum direct bilirubin ≤ 1.5 ULN) (except in subjects with congenital bilirubinemia, such as Gilbert syndrome, direct bilirubinemia ≤ 1.5 ULN)
  * Absolute neutrophil count (ANC) ≥ 1.0 × 109/L
  * Platelet count ≥ 75× 109/L (≥ 50× 109/L if myeloma involvement in the bone marrow is > 50%) and no platelet infusion in the 1 week prior to screening platelet count
  * Creatinine clearance (CrCl) ≥ 30 mL/minute. Creatinine clearance should be calculated using eGFR (Modified Diet in Renal Disese [MDRD])
  * Corrected serum calcium ≤ 13.5 mg/dL (3.4 mmol/L)
  * LVEF ≥ 40%. 2-D transthoracic echocardiogram (ECHO) is the preferred method of evaluation. Multigated Acquisition Scan (MUGA) is acceptable if ECHO is not available.
* Females of childbearing potential (FCBP)* complies with the conditions of the Pregnancy Prevention Plan, including confirmation that she has an adequate level of understanding and must agree to ongoing pregnancy testing and to practice contraception or true abstinence. FCBP must use a highly effective and an additional barrier contraception method simultaneously for 4 weeks before starting therapy, during treatment and dose interruptions and for 5 months after the last dose of study drugs.
* Male subjects must agree to practice contraception if sexually active with FCBP during the treatment and for 5 months after the last dose of study drugs. Males must agree to refrain from donating sperm for at least 90 days after the last dose of carfilzomib and for at least 5 months after the last dose of isatuximab.
* *Note 1: a FCBP is a woman who:
* has achieved menarche at some time point,
* has not undergone a hysterectomy or bilateral oophorectomy or,
* has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).
* Note 2: true abstinence is acceptable when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Previous treatment with anti-myeloma therapy (does not include radiotherapy, biphosphonates, or a single short course of steroid ≤ to the equivalent of dexamethasone 40 mg/day for 4 days).
* Patients with non-secretory MM unless serum free light chains are present and the ratio is abnormal or a plasmacytoma with minimum largest diameters of > 2 cm.
* Patients with plasma cell leukemia, amyloidosis, Waldenstrom Disease, POEMS syndrome
* Meningeal involvement of multiple myeloma
* Patient ineligible for autologous transplantation
* Pregnant or lactating females
* Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to randomization
* Known human immunodeficiency virus infection (HIV)
* Active hepatitis A, B or C infection. Hepatitis C infection (subjects with hepatitis C that achieve a sustained virologic response after antiviral therapy are allowed), or hepatitis B infection (subjects with hepatitis B surface antigen or core antibody that achieve sustained virologic response with antiviral therapy are allowed). Tests to be performed if required per local country regulations. In fact it is not possible to avoid the risk of virological reactivation with the study treatments.
* Unstable angina or myocardial infarction within 4 months prior to randomization, NYHA Class III or IV heart failure, uncontrolled angina, uncontrolled hypertension, (Uncontrolled hypertension, defined as an average systolic blood pressure ≥ 160 mmHg or diastolic ≥ 100 mmHg despite optimal treatment (measured following European Society of Hypertension/European Society of Cardiology 2013 guidelines), pulmonary embolia, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker
* Non-hematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
* Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to randomization as defined by National Cancer Institute Common Toxicity Criteria (NCI CTCAE) 5.0
* Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib) and to PS80; prior hypersensitivity to sucrose, histidine (as base and hydrochloride salt), or any of the components (active substance or excipients) of study treatments that are not amenable to premedication with steroids, or H2 blockers, that would prohibit further treatment with these agents.
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
* Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent
* Pregnant or breastfeeding woman or woman who intends to become pregnant during the participation in the study. FCBP unwilling to prevent pregnancy by the use of 2 reliable methods of contraception for ≥4 weeks before the start of study treatment, during treatment (including dose interruptions), and for at least 28 days following discontinuation of study lenalidomide, or 30 days following discontinuation of carfilzomib or for 5 months after discontinuation of isatuximab treatment, whichever occurs last,
* Male participants who disagree to practice true abstinence or disagree to use a condom during sexual contact with a pregnant woman or a FCBP while participating in the study, during dose interruptions, and for at least 28 days following discontinuation of study lenalidomide, or 30 days following discontinuation of carfilzomib, or for 5 months after discontinuation of isatuximab treatment, whichever occurs last, even if he has undergone a successful vasectomy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of MRD negativity after ASCT consolidation treatment by NGS | The end of consolidation, average of 12 months
  The rate of MRD negativity is determined as the proportion of patients with MRD negativity (≥10-5 sensitivity level) after ASCT consolidation treatment using ITT principle. For patients who withdraw from the study or are lost to follow up before four post ASCT consolidation cycles, the best MRD assessment will be considered. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment.

SECONDARY OUTCOMES:
Post induction MRD negativity rate by NGS | The end of induction, average of 4 months
  The rate of MRD negativity after induction is determined as the proportion of patients with MRD negativity (≥10-5 sensitivity level, NGS) after the induction phase using ITT principle. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment/sample not adequate.
Progression-free survival (PFS) in the 2 arms | approximately up to 5 years
  PFS will be measured from the date of randomization to the date of first observation of PD, or death from any cause as an event. Subjects who have not progressed or who withdraw from the study will be censored at the time of the last complete disease assessment. All subjects who were lost to FU will also be censored at the time of last complete disease assessment
Post light-consolidation MRD negativity rate by NGS | At the end of light-consolidation, average of 24 months
  The rate of MRD negativity after light consolidation is determined as the proportion of patients with MRD negativity (≥10-5 sensitivity level, NGS) after light consolidation phase using ITT principle. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment/sample not adequate. Patients who withdraw from the study or are lost to follow up before MRD evaluation, the best MRD assessment will be considered
Overall Response Rate (ORR) post-induction | Approx 4 months
  Response rate (sCR, CR, VGPR, PR, ORR) will be evaluated according to IMWG Response criteria after induction.
Overall Response Rate (ORR) post-transplant | Approximately 8 months
  Response rate (sCR, CR, VGPR, PR, ORR) will be evaluated according to IMWG Response criteria after ASCT.
Overall Response Rate (ORR) post-consolidation | Approximately 12 months
  Response rate (sCR, CR, VGPR, PR, ORR) will be evaluated according to IMWG Response criteria after consolidation.
Overall Response Rate (ORR) post light-consolidation | Approximately 24 months
  Response rate (sCR, CR, VGPR, PR, ORR) will be evaluated according to IMWG Response criteria after light consolidation.
Post ASCT MRD negativity rate by NGS | After ASCT, approximately 8 months.
  The rate of MRD negativity after ASCT is determined as the proportion of patients with MRD negativity (≥10-5 sensitivity level), NGS using ITT principle. For patients who withdraw from the study or are lost to follow up before ASCT, the best MRD assessment will be considered. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment.
MRD negativity rate by NGF post induction | Approximately 4 months
  The rate of MRD negativity (by NGF) after induction is determined as the proportion of patients with MRD negativity (≥10-5 sensitivity level) after the specific phase using ITT principle. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment. Patients who withdraw from the study or are lost to follow up before MRD evaluation phase, the best MRD assessment will be considered.
MRD negativity rate by NGF post induction | Approximately 8 months
  The rate of MRD negativity (by NGF) after ASCT is determined as the proportion of patients with MRD negativity (≥10-5 sensitivity level) after the specific phase using ITT principle. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment. Patients who withdraw from the study or are lost to follow up before MRD evaluation phase, the best MRD assessment will be considered.
MRD negativity rate by NGF post consolidation | Approximately 8 months
  The rate of MRD negativity (by NGF) after consolidation is determined as the proportion of patients with MRD negativity (≥10-5 sensitivity level) after the specific phase using ITT principle. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment. Patients who withdraw from the study or are lost to follow up before MRD evaluation phase, the best MRD assessment will be considered.
MRD negativity rate by NGF post light consolidation | Approximately 24 months
  The rate of MRD negativity (by NGF) after light consolidation are determined as the proportion of patients with MRD negativity (≥10-5 sensitivity level) after the specific phase using ITT principle. Patients will be classified as MRD positive if they have only MRD positive test results or do not undergo MRD assessment. Patients who withdraw from the study or are lost to follow up before MRD evaluation phase, the best MRD assessment will be considered.
Duration of response | approximately up to 9 years
  Duration of response is defined as the time between first documentation of response (achievement of at least a PR) and PD with deaths owning to causes other than progression not counted, but censored. Responders without disease progression at the cut-off date of final analysis will be censored either at the time of lost to FU, at the time of death due to other cause than PD, or at the at the time of last contact
Duration of MRD negativity (by NGS and NGF) | approximately up to 9 years
  The duration of MRD Negativity (by NGS and NGF) is defined as time between first MRD Negativity and first MRD positivity. Patients without MRD positivity will be censored at last complete assessment
Determine the rate of sustained for 1-year MRD negativity (by NGF and NGS) from post ASCT consolidation to post light consolidation | approximately up to 9 years
  Rate of 1 year sustained MRD negativity by NGS (from post ASCT consolidation to post light consolidation) will be also evaluated.
Determine the time to progression (TTP) | approximately up to 9 years
  From the date of randomization to the date of first disease progression or death per PD, whichever occurs first
Overall Survival (OS) | approximately up to 9 years
  Overall Survival (OS), measured from the date of from randomization to the date the subject's death
Time to next therapy (TNT) | approximately up to 9 years
  TNT will be measured from the date of randomization to the date of next anti-myeloma therapy. Death due to any cause before starting therapy will be considered an event. Subjects who have not progressed or who withdraw from the study will be censored at the time of the last complete disease assessment. Subjects lost to FU will also be censored at the time of last contact.
Progression-free survival on the next line of therapy (PFS2) | approximately up to 9 years
  Progression-free survival on the next line of therapy (PFS2) is defined as the time from randomization to progression on the next line of treatment or death, whichever comes first.

CONTACTS AND LOCATIONS:
Locations (41):
- Het Ziekenhuisnetwerk Antwerpen - Department of Hematology, Antwerp, Belgium
- Czechia (4):
  - Fakultni Nemocnice Brno - Internal Hematology and Oncology Clinic, Brno
  - Fakultni Nemocnice Hradec Kralove - 4th Department of Internal Medicine, Nový Hradec Králové
  - Fakultni Nemocnice Ostrava - Department of Haematooncology, Ostrava
  - Vseobecna Fakultni Nemocnice V Praze - Internal Medicine, Hematology Clinic, Prague
- Germany (3):
  - Medical Center - University Of Freiburg - Department Innere Medizin Klinik für Innere Medizin I, Freiburg im Breisgau
  - University Medical Center Hamburg-Eppendorf - Medizinische Klinik und Polikllinik Onkologie und Knochenmarktransplantation, Haematologie, Hamburg
  - Klinikum rechts der Isar der TU Muenchen AöR - Innere Medizin III-Haematologie/Onkologie, München
- Greece (2):
  - Alexandra Hospital - Department of Clinical Therapeutics National & Kapodistrian University of Athens School of Medicine, Athens
  - Theageneio General Hospital - Department of Hematology Oncology, Thessaloniki
- Italy (11):
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I G M Lancisi G Salesi-SOD Clinica Ematologica, Ancona
  - University Hospital Consorziale Policlinico-U.O. di Ematologia con Trapianto, Bari
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS Istituto Di Ricerca E Di Cura A Carattere Scientifico - U.O. di Ematologia, Bologna
  - Azienda Socio Sanitaria Territoriale Degli Spedali Civili Di Brescia - UOC Ematologia, Brescia
  - Azienda Ospedaliera Santa Croce E Carle - S.C. Ematologia, Cuneo
  - Careggi University Hospital - SOD Ematologia, Florence
  - Azienda Ospedaliero-Universitaria Maggiore Della Carita - SDCU Ematologia, Novara
  - Fondazione IRCCS Policlinico San Matteo-UOC Ematologia 1, Pavia
  - Azienda Sanitaria Locale Di Pescara - U.O. Ematologia, Pescara
  - A.O.U. Città della Salute e della Scienza di Torino-U.O. Ematologia, Torino
  - Azienda Sanitaria Universitaria Giuliano Isontina-SC U.O.C Ematologia, Trieste
- Netherlands (11):
  - Noordwest Ziekenhuisgroep Stichting - Internal Medicine - Hematology, Alkmaar
  - Meander Medisch Centrum -Internal Medicine - Hematology, Amersfoort
  - Amsterdam-Vrije Universiteit Medical Center (VUMC), Amsterdam
  - Amphia Hospital-Internal Medicine - Hematology, Breda
  - Albert Schweitzerplaats 25, Dordrecht
  - Zuyderland Medisch Centrum Stichting - Internal Medicine - Hematology, Geleen
  - Universitair Medisch Centrum Groningen-Department of Haematology, Groningen
  - Medisch Centrum Leeuwarden B.V. - Oncologisch Centrum Leeuwarden (OCL) and Internal Medicine - Hematology, Leeuwarden
  - Sint Antonius Ziekenhuis Stichting-Internal Medicine - Hematology, Nieuwegein
  - ErasmusMC, Rotterdam-Department of Hematology, Rotterdam
  - Haga Hospital - Internal Medicine - Hematology, s-Gravenweg
- Norway (2):
  - Oslo University Hospital HF - Oslo myelomatosesenter, Oslo
  - St. Olavs Hospital HF - Department of Hematology, Trondheim
- Spain (7):
  - Hospital Germans Trias I Pujol - Hematology Service ICO Badalona Clinic, Badalona
  - Hospital Clinic De Barcelona - Myeloma and Amyloidosis Unit, Barcelona
  - Hospital Universitario 12 De Octubre - Hematology, Madrid
  - Hospital Universitario 12 De Octubre -Hematology and Hemotherapy Service, Madrid
  - Clinica Universidad De Navarra - Central Clinical Trials Unit, Pamplona
  - Hospital Universitario De Salamanca-Department of Hematology of the Salamanca University Care Complex, Salamanca
  - Hospital Universitario Marques De Valdecilla -Hematology and Hemotherapy Service, Santander

IPD SHARING:
Plan to Share IPD: Undecided